CLINICAL TRIAL: NCT05396443
Title: A Telehealth Lifestyle Intervention for Black Adolescent Girls at Risk for Type 2 Diabetes: A Pilot Study
Brief Title: Telehealth Lifestyle Program for Black Adolescent Girls at Risk for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-04023546; 1R21MD016986-01 (NIH)
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Childhood; Type2Diabetes
Keywords: Adolescents; Telehealth Lifestyle Program; Diabetes prevention; Black girls; Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Adolescents-Caregiver Dyads (Experimental): Adolescent-caregiver dyads receive 12 week telehealth lifestyle program consisting of a Wellness session, Cooking Experience, and Dance Classes.
  Interventions: Behavioral: Black Girls for Wellness Telehealth

INTERVENTIONS:
Behavioral: Black Girls for Wellness Telehealth — Weekly for 12 weeks, adolescent-caregiver dyads will attend 1) a live stream group Wellness (mindfulness, nutrition lesson, dance class, program reflection) session (90 min/wk) and 2) a home cooking experience using ingredients sent to participants' homes (60 min/wk) with their caregiver. Others in the home (e.g., siblings) will be encouraged to participate in activities as well.

SUMMARY:
The aim of this study is to look at changes in diabetes-related risk factors in Black adolescent girls who are at risk for type 2 diabetes and their primary female caregiver after both participating in a 12-week telehealth lifestyle program.

DETAILED DESCRIPTION:
Enrolled adolescent/caregiver dyads will participate in the 12-week program. Each week, participants will engage in 2 activities: a live virtual Wellness Session and an at-home cooking experience using ingredients sent to them via grocery delivery service.

The study will examine the pre-post difference in overall diet quality, dermal carotenoid levels, physical activity, body composition, and glycemic measures among at-risk black adolescent girls and their caregivers. Investigators hypothesize that after the program, participants' diets will be higher in quality than before.

ELIGIBILITY:
Inclusion Criteria for adolescent participants:

* 12-18 years of age
* self-identify as Black or African American
* have obesity

Exclusion Criteria of adolescent participants:

* pregnant or within 3 months postpartum.
* participated in a formal weight management program within 6 months prior to study.
* currently taking medications or diagnosed with a condition known to influence metabolism, physical activity ability, or cognitive function.
* have previously undergone bariatric surgery.
* have type 2 diabetes.
* unable to speak English or have developmental conditions that interfere with ability to communicate.

Inclusion criteria of caregiver participants:

* 18 years or older.
* proficiency in speaking English.
* live in the same household as the adolescent who will also be enrolled
* prepares the majority (>50%) of meals in the household

Exclusion Criteria of caregiver participants:

* pregnant or within 3 months postpartum.
* unable to speak English or have developmental conditions that interfere with ability to communicate.

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Change in diet quality of adolescent participants, as measured by the Healthy Eating Index Scores | Baseline, 12 weeks [end of study]
  Scores are calculated from three 24-hour diet records, range from 0-100. Higher score reflects that higher alignment between one's diet and dietary recommendations from the Dietary Guidelines for Americans.

SECONDARY OUTCOMES:
Change in dermal carotenoids level | Baseline, 12 weeks [end of study]
  Scores are measured using the Veggie Meter device, range from 0-800. Higher score acts as proxy for fruits and vegetables consumption.
Change in percent time sedentary | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent on sedentary will be calculated.
Change in percent time spent in light activity | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent in light activity will be calculated.
Change in percent time spent in moderate to vigorous activity | Baseline, 12 weeks [end of study]
  Accelerometry data will be collected from wrist accelerometers worn by participants for 7 days. Percent time spent in moderate and vigorous activity will be calculated.
Change in glucose levels | Baseline, 12 weeks [end of study]
  Fasting glucose and 2 hour glucose levels will be collected through an oral glucose tolerance test.
  Subjects enrolled after May 13 2024 will not complete this test to address recruitment barriers (e.g., availability/ time needed for 2 hour test).
Change in fasting insulin levels | Baseline, 12 weeks [end of study]
  Insulin level will be assessed through blood draws on fasting participants.
  Subjects enrolled after May 13 2024 will not be required to fast for this test to address recruitment barriers (e.g., availability for morning appointment) and reduce participant burden.
Change in HbA1c | Baseline, 12 weeks [end of study]
  HbA1c will be assessed through blood draws on fasting participants.
  Subjects enrolled after May 13 2024 will not be required to fast for this test to address recruitment barriers (e.g., availability for morning appointment) and reduce participant burden.
Change in lipid profile | Baseline, 12 weeks [end of study]
  Total, high-density, low-density cholesterol, and triglycerides will be assessed through blood draws on fasting participants.
  Subjects enrolled after May 13 2024 will not be required to fast for this test to address recruitment barriers (e.g., availability for morning appointment) and reduce participant burden.
Change in body mass index | Baseline, 12 weeks [end of study]
  Height will be measured using a stadiometer to the nearest decimal point in cm. Weight will be measured using a scale to the nearest decimal in kg. Body mass index will be calculated using kg/m^2.
Change in body fat percentage | Baseline, 12 weeks [end of study]
  Body fat percentage will be measured using a scale to the nearest decimal.
Change in waist circumference | Baseline, 12 weeks [end of study]
  Waist circumference will be measured using a waist circumference tape to the nearest decimal in cm.
Change in high blood pressure status | Baseline, 12 weeks [end of study]
  Blood pressure will be measured using blood pressure monitors. High blood pressure is considered as reading of >=120/80.

CONTACTS AND LOCATIONS:
Overall Officials: Tashara M Leak, PhD, RD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Brooklyn Methodist Hospital, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT05396443/ICF_000.pdf